CLINICAL TRIAL: NCT00629317
Title: A Randomized, Double-Blind, Placebo-Controlled Trial of Methyl Aminolevulinate + Aktilite in Patients With Facial Photodamage
Brief Title: Trial of Methyl Aminolevulinate Plus Aktilite in Facial Photodamage
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Collaborators: Galderma R&D (Industry)
Responsible Party: Gloria Sanclemente, MD, MSc., Universidad de Antioquia
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: PISUI 2007-031
Record Dates: First submitted 2008-02-25; First posted 2008-03-06 (Estimated); Last update posted 2009-03-16 (Estimated); Status verified 2009-03

CONDITIONS: Skin Aging
Keywords: Skin Aging; Rejuvenation; Photodynamic Therapy; Methyl Aminolevulinate
MeSH Terms: interventions — cetyl alcohol, propylene glycol, sodium lauryl sulfate non-lipid cleansing lotion; methyl 5-aminolevulinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Methyl Aminolevulinate
- B (Placebo Comparator)
  Interventions: Other: Moisturizer

INTERVENTIONS:
Other: Moisturizer — Cetaphil cream(For 3 hours) + Aktilite ( Photodynamic Therapy for 8 minutes)
  Other Names: Cetaphil
  Arms: B
Drug: Methyl Aminolevulinate — Methyl Aminolevulinate cream for 3 hours before Photodynamic therapy ( Aktilite)
  Other Names: Metvix
  Arms: A

SUMMARY:
The aim of the study is to determine the efficacy of MAL + Aktilite versus placebo + Aktilite in facial photodamage in a randomized double blind trial.

DETAILED DESCRIPTION:
It has been demonstrated that photodamage leads to wrinkles, mottled pigmentation, lentigines, telangiectasias, and textural changes, but more importantly, it can also lead to pre-cancerous conditions with the development of actinic keratosis (AK). The majority of photorejuvenation or photodamaged published studies have used 5-Amino-Levulinic acid (5-ALA) as a photosensitizer, and either a blue light or an Intense Pulsed Light source with a 70%-95% global facial skin improvement. The molecular mechanism of such improvement is unknown, but activation of a non-specific immune response in addition to increased fibrosis and new collagen formation, have both been suggested.

Methyl Aminolevulinate ( MAL) is another marketed photosensitizer mainly utilized in Europe. Lipophilicity, higher penetration depth and tumor selectivity has been advocated for MAL compared to 5-ALA. However, its effect in photodamaged skin has not been well documented.

The aim of the study is to determine the efficacy of MAL + Aktilite (PDT) in facial photodamage.

Study Type: Interventional

Study Design: Randomized, double-Blind, placebo-controlled trial. Official Title: A randomized, double-Blind, placebo-controlled trial of Methyl Aminolevulinate + Aktilite in patients with facial photodamage.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects older than 35 years of age and less than 75 years of age
* Subjects with a photodamage grade of 2 or 3 according to a modified Dover´s Global photodamage scale
* Subjects willing to participate according to protocol requirements.
* Patients with signed Informed Consent
* Patients with no exclusion criteria

Exclusion Criteria:

* Pregnant or nursing females.
* Subjects with suspected porphyria, Systemic or cutaneous erythematosus lupus, or any other photosensitizing disorder or drug induced photosensitization.
* Any active infectious skin disorder ( Herpes simplex, molluscum contagiosum, facial warts )
* Subjects with less than 6 months of previous rejuvenation interfering treatments
* Subjects requiring concurrent treatment that would interfere with study objectives and/or assessments.

Ages: 35 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2008-02; Primary Completion 2009-01 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Efficacy in facial global photodamage | 8 months

SECONDARY OUTCOMES:
Facial fine lines, mottled pigmentation, tactile roughness, sallowness, erythema, telangiectasia | 12 months
Histological effect of MAL+PDT in fibrosis and new collagen formation | 12 months
Safety and tolerance | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Sanclemente, Dr, Principal Investigator — Coordinator Group of Investigative Dermatology-GRID; Hector I Garcia, Dr., Study Chair — Coordinator GRAEPIC
Locations (1):
- IPS Universitaria - Universidad de Antioquia, Medellín, Antioquia, Colombia